CLINICAL TRIAL: NCT04062929
Title: Effectiveness of a Short Physical Activity Program on the Level and Barriers to Physical Activity in Individuals With Coronary Artery Disease.
Brief Title: Short Physical Activity Program in Coronary Artery Disease.
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: BAPAC II
Record Dates: First submitted 2019-07-19; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-06

CONDITIONS: Coronary Artery Disease; Motivation
MeSH Terms: conditions — Coronary Artery Disease | interventions — Behavior Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: The investigators included 32 patients who participated to a monocentric 4-day program for secondary prevention in cardiovascular disease, between January 2017 and October 2018. Participation to the program was on a voluntary basis and individuals were referred by their own physician, cardiac rehabilitation center or spontaneously. Eligibility criteria included age 18 years and older, stable coronary artery disease with appropriate medical certificate of fitness and no current medical conditions affecting sports participation. Patients unable to give written constent, with impaired cognitive functions, chronic motor deficiency or severe medical disorder (other than heart disease) significantly affecting functional abilities and individuals with insufficient information about medical history of documented coronary disease were excluded.
  Interventions: Behavioral: 4-day physical activity program with behavioral intervention

INTERVENTIONS:
Behavioral: 4-day physical activity program with behavioral intervention — Each program included 8-12 patients. During the four days, the participants had 4 collective sessions of educational information on PA and heart disease and 2 one-to-one sessions for promoting personal advice and experience on PA behavior. The participants had 6 sessions of PA and 2 food-counseling sessions.

SUMMARY:
Coronary artery diseases (CAD) are multifactorial diseases which prognosis and risk factors are improved with increased physical activity (PA). Thus, CAD rehabilitation (CR) program is mainly based on recovering sufficient exercise capacity and promoting regular personalized PA associated to modifications in lifestyle habits to improve control of cardiovascular risk factors and health-related quality of life. However, most of patients do not achieve the recommended levels of PA which may be partly due to numerous barriers that hamper the return to a physically active lifestyle. One promising interventions strategy is so-called 'brief interventions' (BI) to increase PA in health care settings used to initiate change for an unhealthy behavior in individuals and consisting in "verbal advice, discussion, negotiation or encouragement, with or without written or other support or follow-up". An 'extended brief intervention' (EBI) is similar but usually lasts more than 30 minutes and is delivered on a one-to-one or group basis and can be composed of multiple brief sessions. However, in CAD patients, the effect of such interventions on PA level and behavior remains unclear, as well as predictor patterns associated with better outcomes.

The investigators aimed to assess the effect of a 4-day PA education program with multiple EBI and exercise on the level and barriers to PA in CAD patients and characterize the profile of participants (barriers to PA) with better outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and older
* stable coronary artery disease with appropriate medical certificate of fitness and no current medical conditions affecting sports participation.

Exclusion Criteria:

* Patients unable to give written constent
* Patients with impaired cognitive functions
* Patients with chronic motor deficiency or severe medical disorder (other than heart disease) significantly affecting functional abilities
* Patients with insufficient information about medical history of documented coronary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who participated to the 4-day program "Séjour tremplin: Activité physique et maladie cardiaque" for secondary prevention in cardiovascular disease, between January 2017 and October 2018
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline BAPAC score at 3 months | Two administrations: at the entry in the program and after 3 months follow-up
  Score on the the BAPAC questionnaire (the barriers to appropriate physical activity in CAD patients questionnaire, total score calculated over 55, with higher scores for higher barriers)

SECONDARY OUTCOMES:
Change from Baseline BAPAC score after the 4-day program | Two administrations: at the entry in the program and at the end of the 4-day program
  Score on the the BAPAC questionnaire (the barriers to appropriate physical activity in CAD patients questionnaire, total score calculated over 55, with higher scores for higher barriers)
Change from Baseline Dijon Physical Activity Score at 3 months | Two administrations: at the entry in the program and after 3 months follow-up
  Score on the the Dijon Physical Activity Score (for quantifying the level of physical activity, score over 30 with higher scores for the most active individuals)
BAPAC sensitivity to change (the barriers to physical activity in CAD patients questionnaire, total score calculated over 55, with higher scores for higher barriers) | Two administrations: at the entry in the program and at the end of the 4-day program; Calculation of the sensitivity to change
  Sensitivity to change of the BAPAC scale is calculated with the effect size (ES) and the standardized response mean (SRM). The minimal clinically important difference (MCID) of BAPAC change is calculated using an anchor-based approach calculating the threshold associated with better improvement on Dijon PAS levels (patient changing from low active [<20/30] to active levels [≥20/30]).
BAPAC sensitivity to change (the barriers to physical activity in CAD patients questionnaire, total score calculated over 55, with higher scores for higher barriers) | Two administrations: at the entry in the program andafter 3 months follow-up
  Sensitivity to change of the BAPAC scale is calculated with the effect size (ES) and the standardized response mean (SRM). The minimal clinically important difference (MCID) of BAPAC change is calculated using an anchor-based approach calculating the threshold associated with better improvement on Dijon PAS levels (patient changing from low active [<20/30] to active levels [≥20/30]).

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No